CLINICAL TRIAL: NCT05386615
Title: Post-Exablate Pregnancy Outcomes Registry Study: Exablate Treatment of Symptomatic Uterine Fibroids
Status: Recruiting | Type: Observational
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: UF036
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Uterine Fibroid
Keywords: Uterine Fibroids; Exablate
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Exablate: Observational study of Exablate treatment.
  Interventions: Device: Body System - Functional

INTERVENTIONS:
Device: Body System - Functional — MR-Guided Focused Ultrasound

SUMMARY:
The goal of this Registry Study is to capture clinical pregnancy outcomes and fibroid treatment background data for any subject post-Exablate treatment for their symptomatic fibroids.

DETAILED DESCRIPTION:
This is an observational study only for all consented subjects who undergo an Exablate treatment. The Exablate procedure is a commercial treatment. The objective of this registry is to collect data about the effect of Exablate treatment on potential pregnancy occurrences in this population for two years post-treatment for purposes of labeling updates and overall safety data collection.

ELIGIBILITY:
Inclusion Criteria: - - Eligibility is as per the symptomatic fibroids device indication. - All registry-consented patients following the treatment of their fibroid(s) with the Exablate system. Exclusion Criteria: -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pre- and peri- menopausal women
Study Population: pre- and peri- menopausal women with Uterine Fibroids
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | Through study completion, an average of 2 years.
  All adverse events and/or serious adverse events will be documented and reported according to protocol.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Mayo Clinic, Rochester, Minnesota
- China (3):
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Shanghai No. 1 Hospital, Shanghai
  - Shanghai No.1 Hospital, Shanghai